CLINICAL TRIAL: NCT02534727
Title: Sputum Pharmacokinetics of TB Drugs and Bacterial Drug Resistance
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150187; 15-I-0187
Record Dates: First submitted 2015-08-26; First posted 2015-08-28 (Estimated); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Tuberculosis; Non-Tuberculosis Mycobacteria
Keywords: Pharmacokinetic-Moedeling; Tuberculosis; Therapeutic Drug Monitoring; Drug-Levels; Caseum; Natural History
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Sputum and blood participants: These participants will contribute both blood and sputum to the study
- Sputum only participants: These participants will only contribute sputum to the study

SUMMARY:
Background:

Many people around the world get tuberculosis (TB) and non-tuberculous mycobacteria (NTM) infections. Sometimes medicine that treats these infections does not get to where the bacteria are in the lungs. Researchers want to find a way to tell if enough medicine is getting to where it is needed in the lungs. They will look at how much medicine is in your sputum (what you cough up) compared to how much is in your blood. They will also investigate a new test to quickly figure out what medicines are likely to treat TB effectively.

Objective:

To determine the relationship between the concentration of TB drugs in plasma and sputum over time.

Eligibility:

People ages 18 and older who have TB or NTM infection that is suspected to be drug resistant. They must be taking TB or NTM medicines.

Design:

Participants will be screened with medical history.

Participants will be in the study for 2 8 days.

Participants will give 3 or more sputum samples over at least 2 different days. They will cough sputum into a cup.

Participants will have blood drawn 4 times a day on 2 different days.

DETAILED DESCRIPTION:
This study will support two avenues of research, pharmacokinetics (PK) of drugs used to treat tuberculosis and resistance to those drugs that has been developed by the pathogen. Given the high inter-individual variability in TB drug exposure, therapeutic drug monitoring would be of value to adjust the drug dose in TB patients in order to improve clinical outcome and minimize toxicity. It is not practiced in most settings for reasons associated with costs but also because blood collection is an invasive procedure. Sputum on the other hand is often produced spontaneously and discarded as waste. Drug levels can be measured in sputum just as in plasma. Here we will test the hypothesis that sputum drug levels are predictive of drug concentrations in plasma and/or in specific lesion compartments such as the caseum of open cavities. We will also characterize the exposure of standard 1st and 2nd line TB drugs at one of the sites of infection, since sputum is in direct contact with cavity caseum. The subjects will contribute three or more sputum samples spontaneously produced over at least two days and four blood samples following drug administration on two different days (8 blood samples total). The data will be analyzed using population PK modeling approaches to generate concentration-time profiles and 24-hour area under the curve (AUC) of each study drug in sputum. Correlations between these values, plasma and lesion AUCs will be examined. We will draw from a recently completed TB lesion pharmacokinetic study (www.ClinicalTrials.gov #NCT00816426) to seek correlations between drug exposure in sputum and in pulmonary lesions. In addition to drug concentrations, sputum will be cultured by standard methods to isolate Mycobacterium tuberculosis (Mtb), determine the drug resistance profile, and be saved for testing a second generation of the Xpert TB XDR assay.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. At least 18 years of age
  2. Diagnosis of TB (and/or NTM for NIH clinical center subjects)
  3. Ongoing signs and/or symptoms of pulmonary TB (and/or NTM at the NIH CC)
  4. Suspected drug resistance (drug susceptible allowed at the NIH CC)
  5. Available to provide at least 3 sputa over 2 or more days
  6. Taking anti-tuberculosis medicines (or NTM meds at NIH CC) during the time sputa are provided
  7. Thought likely to be Mycobacterium culture positive (including NTM infected for the NIH CC) by enrolling physician
  8. GeneXpert MTB/RIF sputum TBpositive (China subjects only)
  9. Likely able to produce sputum samples while on study
  10. Willing to provide blood samples
  11. Willing to have samples stored

EXCLUSION CRITERIA:

1. Acute liver or kidney disease
2. Conditions which compromise the subject s ability to take or absorb oral drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective trial of the pharmacokinetics of TB drugs in the sputum and blood of drug susceptible and drug resistant subjects at the Henan Provincial Chest Hospital in Zhengzhou, China and at the NIH Clinical Center in Bethesda, MD. Patients (inpatients or outpatients) being treated for TB (including those with NTM at the NIH CC) were asked to join the study.@@@@@@@@@@@@
Sampling Method: Non-Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2016-01-27 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the AUC (0-24) in sputum and blood. | 0-24 hrs
  drug-specific correlation coefficients of the AUCs for sputum and blood

SECONDARY OUTCOMES:
drug-specific time-concentration curves, as well as drug exposure in sputum relative to that in cavity caseum | Throughout
  Estimation of time-concentration curves, as well as variance components of sputum PK parameters to better inform sputum PK sampling in future studies. Additionally, the relationship between drug-specific exposures in cavity caseum, from historical data, and that in sputum will be evaluated using correlation coefficients.

CONTACTS AND LOCATIONS:
Overall Officials: Clifton E Barry, Ph.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (2):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States
- Henan Provincial Chest Hospital, Zhengzhou, China

REFERENCES:
- [Background] Wilkins JJ, Savic RM, Karlsson MO, Langdon G, McIlleron H, Pillai G, Smith PJ, Simonsson US. Population pharmacokinetics of rifampin in pulmonary tuberculosis patients, including a semimechanistic model to describe variable absorption. Antimicrob Agents Chemother. 2008 Jun;52(6):2138-48. doi: 10.1128/AAC.00461-07. Epub 2008 Apr 7. PMID 18391026
- [Background] Dartois V. Drug forgiveness and interpatient pharmacokinetic variability in tuberculosis. J Infect Dis. 2011 Dec 15;204(12):1827-9. doi: 10.1093/infdis/jir662. Epub 2011 Oct 21. No abstract available. PMID 22021619
- [Background] Peloquin C. Use of therapeutic drug monitoring in tuberculosis patients. Chest. 2004 Dec;126(6):1722-4. doi: 10.1378/chest.126.6.1722. No abstract available. PMID 15596662
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-I-0187.html